CLINICAL TRIAL: NCT02876471
Title: Huai'an First People's Hospital,Nanjing Medical University
Brief Title: Continuous Monitoring Nocturnal Beat-to-beat Blood Pressure Fluctuation in OSA With or Without Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huai'an No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Xu J, Doctor of the sleep center in Huai'an NO.1People's Hospital, Huai'an No.1 People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Huaian1PH
Record Dates: First submitted 2016-08-10; First posted 2016-08-23 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Blood Pressure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSA group (No Intervention): 100 severe OSA patients without hypertension were enrolled. Primal evaluations including office blood pressure, Epworth sleepiness scale score(ESS),demographic and anthropometric data The full night polysomnogram was performed, recording nocturnal blood pressure, oximetry, beat-to-beat BPV, AHI, BP event was calculated
- OSA with hypertension (Other): 100 severe OSA patients with hypertension were enrolled. Primal evaluations including office blood pressure, Epworth sleepiness scale score(ESS), antihypertensive medicine demographic and anthropometric data. The full night polysomnogram was performed, recording nocturnal blood pressure, oximetry, beat-to-beat BPV, AHI, BP event was calculated.Screening of 40 newly diagnosed patients with hypertension and subjects with poor blood pressure control, the investigators would give one-night CPAP.
  Interventions: Other: CPAP

INTERVENTIONS:
Other: CPAP — OSA complicated with hypertension：In order to avoid the effects of drugs on this study, we calculated the time to stop based on the half-life of patients taking oral drugs and last time administration time. The subject who withdrawal time was less than three days was enrolled in our study. These patients were hospitalized and close monitoring of blood pressure, for blood pressure three times greater than 180/110mmHg or appearing dizziness, headache and other clinical syndrome, we give a timely clinical intervention and get rid of our study. Screening of 40 newly diagnosed patients with hypertension and subjects with poor blood control,the investigators would give one-night CPAP
  Arms: OSA with hypertension

SUMMARY:
Emerging evidence suggests that there is a causal link between obstructive sleep apnea(OSA) and hypertension. Patient with this syndrome exhibit several characteristics: high prevalence, frequent non-dipper status, diastolic and nocturnal predominance, which are related to clinical and subclinical organ damage in heart and brain. However, the influence of OSA on nocturnal hypertension development has not yet been clarified. Blood pressure variability (BPV) plays a role in vascular damage, independent of blood pressure. Apnea overloads the autonomic cardiovascular control system and may influence BPV,which is classified by different time interval, including beat-to-beat, hour-to-hour day-to-night changes or long-term, for example days, weeks, months, seasons, and even years. All BPV abnormalities are associated with an increased incidence of cardiovascular events and mortality. The investigators pre-experiment estimate BPV by ambulatory blood pressure monitoring (ABPM), which unable to capture the BP fluctuation accurately during the apnea event. The small studies exam beat-to-beat BP and OSA，and the investigators can't couple the events with blood fluctuation, also incapable calculate the correlation of them. This study is aimed to use pulse transmit time(PTT) based blood pressure measurement which can be useful for continuous monitoring of blood pressure to monitor nocturnal beat-to-beat blood pressure fluctuation in OSA with or without hypertension, investigating the degree of relevance between hypoxia, AHI, nocturnal hypertension development and BPV. Besides that the investigators also evaluate the effect of continuous positive airway pressure(CPAP) on blood pressure and nocturnal beat-to-beat BPV.

DETAILED DESCRIPTION:
Methods:

Between March 2016 and December 2016,the investigators initially recruited 450 individuals reporting severe habitual snoring. Primal evaluations including office blood pressure, Epworth Sleepiness Scale Score(ESS), antihypertensive medicine demographic and anthropometric data. Then overnight polysomnography were performed. Of them,100 were severe OSA (AHI>30 episode/h) with hypertension, who were agreed to stop taking antihypertensive medicine. The investigators calculated the time to stop based on the half-life of patients taking oral drugs and last time administration time. The subject who withdrawal time was less than three days was enrolled in this study. These patients were hospitalized and close monitoring of blood pressure, for blood pressure three times greater than 180/110mmHg or appearing dizziness, headache and other clinical syndrome, the investigators will give a timely clinical intervention and get rid of this study. The control group consisted of 100 subjects just with severe OSA whose blood pressure is normal. The investigators recorded nocturnal blood pressure, oximetry, beat-to-beat BPV, AHI, BP event was calculated. Screening of 40 newly diagnosed patients with hypertension and subjects with poor blood pressure control, the investigators would give one-night continuous positive airway pressure(CPAP) to compare the AHI, the mean nocturnal systolic blood pressure and diastolic blood pressure, the number of blood events before and after short-term CPAP therapy, to compare the AHI, the mean nocturnal systolic blood pressure and diastolic blood pressure, the number of blood events before and after short-term CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* severity OSA (AHI>30 episode/h)
* aged between 18 to 70 yeas
* blood pressure≦180/110mmHg

Exclusion Criteria:

* blood pressure>180/110mmHg
* severe clinical events such as coronary artery disease, heart failure,cerebrovascular disease or renal failure
* diabetes
* patients with suspected secondary hypertension
* patients with pulmonary disease being treated with bronchodilators, corticosteroids, or oxygen
* individuals who are able to perform the test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Office hypertension | 2 hours
  as BP≧140/90mmHg on three different occasions (according to standard guidelines)
nocturnal hypertension | 1 night
  as nighttime systolic blood pressure
  ≧120mmHg and/or70mmHg(diastolic blood pressure)
hypoxemia | 1 night
  as the total time and the number of pulse oxygen less than 90% ,the minimum lowest pulse oxygen saturation during sleep
Beat-to-Beat BPV | 1 night
  as the a increase in systolic blood pressure(SPB) from baseline during an apnea event
BP event | 1 night
  the number of beat-to-beat BPV>10mmHg divided by sleep time
Apnea-hypopnea index(AHI) | 1 night
  AHI was defined as the number of apnea plus hypopnea episode per hour of sleep and was the summary measurement of the occurrence of sleep -disordered breathing.Apnea was defined as a reduction of airflow of at least 90% on the oronasal thermistor for at least 10s(it was considered obstructive if respiratory effort was absent).Hypopneas was scored when the magnitude of the signal decreased by at least 30% of the baseline amplitude of the nasal pressure transducer for at least 10s and was associated with a 4% or greater drop in oxygen saturation,as measured by finger pulse oximetry.
time of event | 1 night
  as the total time of apnea and hypopnea during sleep

CONTACTS AND LOCATIONS:
Overall Officials: Zi Li Meng, Master, Study Chair — Huai'an First People's Hospital
Locations (1):
- Department Of Respiratory Medicine,Huai'an First People's Hospital,Nanjing Medical University, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothwell PM, Howard SC, Dolan E, O'Brien E, Dobson JE, Dahlof B, Sever PS, Poulter NR. Prognostic significance of visit-to-visit variability, maximum systolic blood pressure, and episodic hypertension. Lancet. 2010 Mar 13;375(9718):895-905. doi: 10.1016/S0140-6736(10)60308-X. PMID 20226988
- [Background] Steinhorst AP, Goncalves SC, Oliveira AT, Massierer D, Gus M, Fuchs SC, Moreira LB, Martinez D, Fuchs FD. Influence of sleep apnea severity on blood pressure variability of patients with hypertension. Sleep Breath. 2014 May;18(2):397-401. doi: 10.1007/s11325-013-0899-z. Epub 2013 Oct 3. PMID 24092449
- [Background] Johansson JK, Niiranen TJ, Puukka PJ, Jula AM. Prognostic value of the variability in home-measured blood pressure and heart rate: the Finn-Home Study. Hypertension. 2012 Feb;59(2):212-8. doi: 10.1161/HYPERTENSIONAHA.111.178657. Epub 2012 Jan 3. PMID 22215704
- [Derived] Xu J, Ding N, Chen L, Zhang Y, Huang M, Wang Y, Meng Z, Zhang X. Inducers of post-apneic blood pressure fluctuation monitored by pulse transfer time measurement in obstructive sleep apnea varied with syndrome severity. Sleep Breath. 2019 Sep;23(3):769-776. doi: 10.1007/s11325-018-1770-z. Epub 2019 Jan 12. PMID 30637570
- [Derived] Xu J, Ding N, Zhang X, Wang N, Sun B, Zhang R, Xie X, Wan Z, Gu Y, Zhang S, Hong Y, Huang M, Meng Z. Nocturnal blood pressure fluctuation and associated influential factors in severe obstructive sleep apnea patients with hypertension. Sleep Breath. 2018 Dec;22(4):1045-1052. doi: 10.1007/s11325-018-1634-6. Epub 2018 Mar 9. PMID 29524090